CLINICAL TRIAL: NCT00230776
Title: A 14-Week, Randomized, Double-Blind, Placebo-Controlled Trial Of Pregabalin Twice Daily In Patients With Fibromyalgia
Brief Title: A Controlled Pregabalin Trial In Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081077
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2012-10

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

INTERVENTIONS:
Drug: pregabalin
Drug: placebo

SUMMARY:
To evaluate the efficacy and safety of pregabalin compared with placebo for the relief of pain associated with fibromyalgia and improvement of function of patients with fibromyalgia

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the ACR criteria for fibromyalgia (ie, widespread pain present for at least 3 months, and pain in at least 11 of 18 specific tender point sites.
* Patients must have a score of >40 mm on the Visual Analog Scale

Exclusion Criteria:

* Patients with any widespread inflammatory musculoskeletal disorders, widespread rheumatic diseases other than fibromyalgia, active infections, or untreated endocrine disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740
Dates: Start 2005-10; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of pregabalin for pain relief by comparing the mean pain score between treatment groups and placebo.

SECONDARY OUTCOMES:
To evaluate the efficacy of pregabalin for improvement in sleep, fatigue, health-related quality of life, functioning and mood disturbance associated with fibromyalgia. To evaluate safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (79):
- United States (79):
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Pismo Beach, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Palm Beach Gardens, Florida
  - Pfizer Investigational Site, Palm Harbor, Florida
  - Pfizer Investigational Site, Sunrise, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Gurnee, Illinois
  - Pfizer Investigational Site, Moline, Illinois
  - Pfizer Investigational Site, Morton Grove, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Prairie Village, Kansas
  - Pfizer Investigational Site, Pratt, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Kenner, Louisiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Lansing, Michigan
  - Pfizer Investigational Site, Chaska, Minnesota
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Morristown, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Endwell, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, West Seneca, New York
  - Pfizer Investigational Site, Asheville, North Carolina
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Salisbury, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Minot, North Dakota
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Norristown, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Goose Creek, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Myrtle Beach, South Carolina
  - Pfizer Investigational Site, Summerville, South Carolina
  - Pfizer Investigational Site, Chattanooga, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Milan, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Bedford, Texas
  - Pfizer Investigational Site, Georgetown, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Killeen, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Woodstock, Vermont
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Everett, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Clair A, Emir B. The safety and efficacy of pregabalin for treating subjects with fibromyalgia and moderate or severe baseline widespread pain. Curr Med Res Opin. 2016;32(3):601-9. doi: 10.1185/03007995.2015.1134463. Epub 2016 Jan 27. PMID 26694975
- [Derived] Straube S, Moore RA, Paine J, Derry S, Phillips CJ, Hallier E, McQuay HJ. Interference with work in fibromyalgia: effect of treatment with pregabalin and relation to pain response. BMC Musculoskelet Disord. 2011 Jun 3;12:125. doi: 10.1186/1471-2474-12-125. PMID 21639874
- [Derived] Bhadra P, Petersel D. Medical conditions in fibromyalgia patients and their relationship to pregabalin efficacy: pooled analysis of Phase III clinical trials. Expert Opin Pharmacother. 2010 Dec;11(17):2805-12. doi: 10.1517/14656566.2010.525217. Epub 2010 Nov 2. PMID 21039311
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081077&StudyName=A+Controlled+Pregabalin+Trial+In+Fibromyalgia